CLINICAL TRIAL: NCT02698111
Title: Donafenib Monotherapy for Previously Treated Metastatic Nasopharyngeal Carcinoma：an Open-label,Phase 1 Study.
Brief Title: Donafenib Monotherapy for Previously Treated Metastatic Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate policy adjustments
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGDN1B
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma,donafeinib
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafeinib (Experimental): donafenib 200mg,bid
  Interventions: Drug: Donafenib

INTERVENTIONS:
Drug: Donafenib — donafenib 200mg，bid
  Other Names: CM4307

SUMMARY:
The investigators do the clinical trial (patients with metastatic nasopharyngeal carcinoma treated with donafenib after failure of standard therapy) to assess safety and efficacy of donafenib in patients with metastatic nasopharyngeal carcinoma, progressing after all approved standard therapies.

DETAILED DESCRIPTION:
The study is an open-label, phase 1B study recruiting 18 patients. Patients were eligible to participate when they have histological or cytological documentation of the nasopharyngeal carcinoma. They must have received locally and currently approved standard therapies and to have disease progression after the last administration of the last standard therapy or to have stopped standard therapy because of unacceptable toxic effects. The available standard therapies have to include one or more drugs of the following as were licensed: a fluoropyrimidine,taxane,DDP, gemcitabine.

Patients have to be aged 18 years or older and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; life expectancy of at least 3 months;and adequate bone-marrow, liver, and renal function at the start of the trial. Patients could not participate if they had previously received sorafenib or had uncontrolled medical disorders. All patients receive best supportive care, excluding other investigational antitumour agents or antineoplastic chemotherapy, hormonal therapy, or immunotherapy.Patients receive oral donafenib 200mg (CM4307) of each 4 week cycle until disease progression,death, unacceptable toxic effects, withdrawal of consent by the patient,or decision by the treating physician that discontinuation would be in the patient's best interest.The primary endpoint is safety.The second endpoint is progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological documentationof the nasopharyngeal carcinoma;
* Have received system standard therapies and to have disease progression(RECIST1.1) or to have stopped standard therapy because of unacceptable toxic effects.
* Standard therapies including as many of the following as were licensed: a fluoropyrimidine,taxol,DDP,or gemcitabine;
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Life expectancy of at least 3 months;
* Have adequate bone-marrow, liver, and renal function at the start of the trial. • Prothrombin time international normalized ratio≤2；or prothrombin time≤16 seconds;or activated partial thromboplastin time(APTT) ≤43 seconds;or TT≤21 seconds.

Exclusion Criteria:

* Patients have prior treatment with sorafenib;
* Patients have Central nervous system(CNS) involvement;
* patients have uncontrolled medical disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 2 years
  Percent of adverse events

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  Median of progression of free survival
Response Rate | 1 year
  Percent of patients of PR&CR

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Kai Shi, Doctor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Sciencess
Locations (1):
- Cancer Hospital of Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No